CLINICAL TRIAL: NCT03758456
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess the Safety and Tolerability of HAL-MRE1 Subcutaneous Immunotherapy in Adult Subjects With Ragweed Induced Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma
Brief Title: HAL-MRE1 Subcutaneous Immunotherapy in Ragweed Allergic Patients First-in-human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAL-MRE1/PR0051
Record Dates: First submitted 2018-11-07; First posted 2018-11-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Rhinitis, Allergic; Rhinoconjunctivitis, Allergic
Keywords: Subcutaneous immunotherapy; Ragweed pollen; Allergic rhinitis/rhinoconjunctivitis; Safety; Tolerability
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HAL-MRE1 0 AUeq (Placebo Comparator): 15 subjects will receive placebo. Subjects will receive 7-9 incremental weekly injections. All doses will be subcutaneously injected in a double-blind fashion in the upper arm.
  Interventions: Biological: HAL-MRE1
- HAL-MRE1 5,000 AUeq (Experimental): 10 subjects will receive HAL-MRE1 5,000 AUeq. Subjects will receive 6-8 incremental weekly injections until reaching the maximum dose of 5,000 AUeq. Subsequently, 1 repeated maximum dose injection will be given 1 week later (total treatment period will be approximately 7-9 weeks). All doses will be subcutaneously injected in a double-blind fashion in the upper arm.
  Interventions: Biological: HAL-MRE1
- HAL-MRE1 10,000 AUeq (Experimental): 10 patients will receive HAL-MRE1 10,000 AUeq. Subjects will receive 6-8 incremental weekly injections until reaching the maximum dose of 10,000 AUeq. Subsequently, 1 repeated maximum dose injection will be given 1 week later (total treatment period will be approximately 7-9 weeks). All doses will be subcutaneously injected in a double-blind fashion in the upper arm.
  Interventions: Biological: HAL-MRE1
- HAL-MRE1 20,000 AUeq (Experimental): 10 patients will receive HAL-MRE1 20,000 AUeq. Subjects will receive 6-8 incremental weekly injections until reaching the maximum dose of 20,000 AUeq. Subsequently, 1 repeated maximum dose injection will be given 1 week later (total treatment period will be approximately 7-9 year). All doses will be subcutaneously injected in a double-blind fashion in the upper arm.
  Interventions: Biological: HAL-MRE1

INTERVENTIONS:
Biological: HAL-MRE1 — HAL-MRE1 is a liquid suspension for subcutaneous administration containing aluminum hydroxide adsorbed modified allergens extracted from ragweed pollen.

SUMMARY:
The aim of this first-in-human phase I study is to assess the safety and tolerability of HAL-MRE1 subcutaneous immunotherapy in subjects suffering from ragweed pollen-induced allergic rhinitis/rhinoconjunctivitis with or without asthma.

The study has 4 treatment groups: 1 placebo group and 3 groups treated with different doses of HAL-MRE1.

DETAILED DESCRIPTION:
A chemically modified, aluminum hydroxide adsorbed ragweed extract (HAL-MRE1) for subcutaneous administration was developed for the treatment of ragweed pollen-induced allergic rhinitis/rhinoconjunctivitis (ARC) with or without asthma. The aim of this first-in-human phase I study is to assess the safety and tolerability of HAL-MRE1 subcutaneous immunotherapy in subjects suffering from ragweed pollen-induced ARC with or without asthma.

The study will consist of 3 staggered cohorts of 15 subjects each who are randomly assigned to the active or placebo group in a 2:1 manner using block randomization.

A one month gap must be maintained between the end of the ragweed pollen peak season (2018) and subject randomization into the study. The study has seasonal constraints; subjects with concomitant tree and/or grass pollen allergies must complete study treatment before any allergy symptoms due to tree and/or grass pollen exposure develop or start study treatment after the symptoms caused by the tree and/or grass pollen exposure have disappeared.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female subjects aged ≥18 and ≤65 years.
3. Documented diagnosis of allergic rhinitis/rhinoconjunctivitis (ARC) to ragweed pollen. A documented diagnosis is a documented medical history of ARC symptoms that required treatment after ragweed pollen exposure. Subjects experienced allergy symptoms that required treatment during the previous 2 ragweed seasons, with or without concomitant asthma (asthma must be controlled).
4. Positive nasal provocation test for ragweed pollen at screening or within the last 6 months.
5. Positive skin prick test to ragweed allergen at screening or within the last 6 months.
6. Positive serum specific IgE test for ragweed allergen (IgE level ≥0.7 U/mL).
7. Forced expiratory volume >70 % or peak expiratory flow >80 % of predicted value.
8. For asthmatic subjects: asthma control test (ACT) score ≥20.
9. Subjects are capable and willing to maintain a log of adverse events and concomitant medication throughout the study, as well as to complete a diary 24 hours post investigational medical product injection.
10. Negative pregnancy test at screening for females of childbearing potential.
11. Females of childbearing age must be using an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study. Contraceptive measures considered adequate are:

    1. hormonal contraceptives such as contraceptive pills, transdermal patches, intrauterine devices, intrauterine system implants, or vaginal rings (started at least 4 weeks prior to investigational medical product administration).
    2. double barrier methods e.g. condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent.
    3. sterilization (male or female).
    4. participants who are postmenopausal (12 consecutive months without a period) for at least 2 years.
    5. sexual abstinence or having no sexual relationship with a man.

Exclusion Criteria:

1. History of anaphylaxis with cardio respiratory symptoms (food allergy, venom allergy, drugs or/and idiopathic reaction).
2. Alcohol, drug or medication abuse in the past.
3. Any clinically significant abnormal laboratory parameter at screening as per investigator's discretion.
4. Clinically relevant sensitization to other allergens if clinical symptoms are expected during the study.
5. Uncontrolled asthma.
6. Participation in a clinical interventional study within the last 3 months (e.g. new investigational drug or biological), or plans to participate in another clinical trial during this study, or participation in an observational study (e.g. post marketing study) within the last 30 days unless the observational study aimed to investigate the intradermal test.
7. Subjects who received immunotherapy for any specific allergen 3 years prior to screening or during the study period.
8. Subjects who were ever treated with any ragweed allergen specific immunotherapy.
9. Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs.
10. Subjects undergoing any immunosuppressive treatment (including anti-IgE therapy) within the last 6 months prior to inclusion in the study as well as during the study.
11. Active malignancies or any malignant disease during the 5 years prior to screening.
12. Severe uncontrolled diseases that, in the opinion of the investigator, could increase the risk for subjects participating in the study, including but not limited to: any severe or unstable lung diseases; endocrine diseases; clinically significant renal or hepatic diseases, or hematological disorders; or severe ongoing symptomatic allergic diseases.
13. Active or acute inflammation or infection of the target organs (nose, eyes) at screening.
14. Diseases with a contra-indication for the use of adrenaline (e.g. hyperthyroidism, glaucoma).
15. Lactation.
16. Severe psychiatric, psychological, or neurological disorders.
17. Subjects who have any direct working relationship with the (sub-) investigator or study site personnel or are first degree relatives or partners of the investigator or study site personnel or are employees of the sponsor.
18. Known allergy or hypersensitivity to an excipient in the study drug or placebo.
19. Subjects receiving the prohibited previous and concomitant medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Occurence of local and systemic reactions | Through study completion, approximately 10 weeks
  Number, intensity and seriousness of early (within 30 mins from injection), delayed (within 30mins and 3 hours from injection) and late (from 3 hours to 24 hours after injection) local reactions (>8 cm wheal size swelling at injection site) as well as early, delayed and late systemic reactions.

SECONDARY OUTCOMES:
Occurence of other local reactions | Through study completion, approximately 10 weeks
  Number, intensity and seriousness of other local reactions like itching, pain and redness at injection site.
Occurrence of treatment emergent adverse events | Through study completion, approximately of 10 weeks
  Treatment emergent adverse events will be collected by reporting of adverse events and by clinical relevant changes in e.g. laboratory values, vital signs, physical exam, and lung function in plasma and urine
Number of subjects that reach maximum dose | Through study completion, approximately of 10 weeks
  The number of subjects in each cohort who reach the maximum dose is indicative of HAL-MRE1 tolerability.
Number of injections to reach maintenance dose | Through study completion, approximately of 10 weeks
  The number of injections that subjects in each cohort need to reach the maximum dose will provide an indication of HAL-MRE1 tolerability.
Immunoglobulin Levels | Pre-treatment and after the repeated maintenance dose visit (after 8 to 10 weeks)
  Short term pharmacodynamic effects of HAL-MRE1 will be measured by determining the change in serum levels of allergen specific immunoglobulins (IgE, IgG and IgG4) pre- and post-study treatment in the HAL-MRE versus placebo treated groups.
Change in wheal size after skin prick test | Pre-treatment and after the repeated maintenance dose visit (after 8 to 10 weeks)
  Exploratory efficacy data will be obtained by measuring the change in wheal size following skin prick test with ragweed extract pre- and post-treatment in the HAL-MRE1 versus placebo treated groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Inflamax Research Ltd.
Locations (1):
- Inflamax Research Inc., Mississauga, Canada